CLINICAL TRIAL: NCT03515460
Title: Acute Effects of Standardized Oral Carbohydrate and Fat Loads, and the Association of Carbohydrate and Fat Loads, on Systemic Microvascular Endothelial Function in Healthy Individuals.
Brief Title: Acute Effects of Oral Carbohydrate and Fat Loads on Systemic Microvascular Endothelial Function in Healthy Individuals.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Cardiology, Laranjeiras, Brazil (Other Government)
Responsible Party: Principal Investigator, Eduardo Tibirica, MD, PhD, Senior Researcher, MD, PhD, National Institute of Cardiology, Laranjeiras, Brazil
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CAAE 86854318.8.0000.5272
Record Dates: First submitted 2018-04-20; First posted 2018-05-03 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Metabolic Syndrome
Keywords: vascular endothelial function; systemic microvascular reactivity; dysglycemia; dyslipidemia
MeSH Terms: conditions — Metabolic Syndrome; Dyslipidemias | interventions — Diet Therapy; Sugars

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- sugar oral load (Experimental): oral ingestion of a high carbohydrate meal
  Interventions: Other: sugar oral load
- fat oral load (Experimental): oral ingestion of a high fat meal
  Interventions: Other: fat oral load
- sugar and fat oral loads (Experimental): oral ingestion of a high carbohydrate and fat meal
  Interventions: Other: sugar and fat oral load

INTERVENTIONS:
Other: sugar oral load — The individuals will receive a sugar oral load (high sugar meal)
  Other Names: dietary intervention
  Arms: sugar oral load
Other: fat oral load — The individuals will a receive fat oral load (high fat meal)
  Other Names: dietary intervention
  Arms: fat oral load
Other: sugar and fat oral load — The individuals will a receive sugar and fat oral load (high sugar and high fat meal)
  Other Names: dietary intervention
  Arms: sugar and fat oral loads

SUMMARY:
The present study was designed to evaluate vascular endothelial dysfunction resulting from the oral ingestion of high loads of sugar and fat meals in healthy individuals.

DETAILED DESCRIPTION:
The chronic and elevated consumption of fat and carbohydrates is associated with the initiation and the progression of cardiovascular and metabolic diseases, including diabetes, obesity and metabolic syndrome. In general, chronic diseases are related to underlying modifiable cardiovascular risk factors, including high blood pressure, high plasma lipids and glucose, physical inactivity, overweight and obesity, as well as smoking habits.

Vascular endothelial dysfunction is one of the earliest findings in the pathophysiology of atherosclerosis and also an important predictor of cardiovascular events. Moreover, it has already been demonstrated that acute oral ingestion of high loads of sugar and fat meals induces transient vascular endothelial dysfunction, which over time could lead to cardiovascular disease.

Thus, the present study aimed at investigating the individual contributions of sugar and fat ingestion on systemic microvascular endothelial reactivity.

ELIGIBILITY:
Inclusion Criteria:

* healthy individuals presenting body mass index between 18.5 e 24.9 kg/m2

Exclusion Criteria:

* dysglycemia and dyslipidemia
* overweight and obesity

Ages: 20 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2018-12-10 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-20 (Actual)

PRIMARY OUTCOMES:
endothelial-dependent microvascular function | one day
  alterations in skin microvascular conductance using laser-based methods

CONTACTS AND LOCATIONS:
Overall Officials: EDUARDO TIBIRICA, MD, PhD, Principal Investigator — National Institute of Cardiology
Locations (1):
- National Institute of Cardiology, Ministry of Health, Brazil, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: Undecided